CLINICAL TRIAL: NCT03178344
Title: Rational Optimization of tACS for Targeting Thalamo-Cortical Oscillations (Experiment 2)
Brief Title: Effect of tACS Stimulation on Alpha Oscillations
Acronym: AIMS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16-1911a; R01MH111889-01 (NIH)
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Results first posted 2018-12-07 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Each participant will receive sham stimulation or 10 Hz tACS stimulation at two separate sessions. The order will be randomized (ie, half the participants will receive sham stimulation at the first session and 10 Hz tACS stimulation at the second session, and the other half will receive 10 Hz tACS stimulation at the first session and sham stimulation at the second session).
Who Masked: Participant, Investigator
Masking Description: This study will follow a double-blind experimental design, so neither the participant nor the experimenter will know what kind of stimulation the participant is receiving at what session. A separate unblinded monitor, who will not interact with the participants, will be responsible for creating the stimulation codes for each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham Stimulation, then Alpha Stimulation (Experimental): Participants receive sham stimulation at the first session, followed by a 5-9 day washout period and alpha stimulation at the second session.
  Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham.
  Participants will receive 2 mA of alternating current stimulation at a frequency of 10 Hz for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  Interventions: Device: XCSITE100 Stimulator tACS; Device: XCSITE100 Stimulator Sham
- Alpha Stimulation, then Sham Stimulation (Experimental): Participants receive alpha stimulation at the first session, followed by a 5-9 day washout period and sham stimulation at the second session.
  Participants will receive 2 mA of alternating current stimulation at a frequency of 10 Hz for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham.
  Interventions: Device: XCSITE100 Stimulator tACS; Device: XCSITE100 Stimulator Sham

INTERVENTIONS:
Device: XCSITE100 Stimulator tACS — Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
  Other Names: tACS
Device: XCSITE100 Stimulator Sham — The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session.
  Other Names: Sham tACS

SUMMARY:
Transcranial Alternating Current Stimulation (tACS) is one method that has been demonstrated to enhance alpha oscillations in healthy participants by applying weak electrical currents to the scalp to modulate rhythmic brain activity patterns. This study will involve tACS-induced frontal alpha oscillations, EEG recordings, and other physiological and biological measures.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Negative pregnancy test for female participants

Exclusion Criteria:

* History of major neurological or psychiatric illness, including epilepsy
* Medication use associated with neurological or psychiatric illnesses
* Currently undergoing counseling or psychotherapy treatment for depression, anxiety, eating disorders, PTSD or other behavioral conditions
* First degree relative (parent, sibling, child) with major neurological or psychiatric illness
* Prior brain surgery
* Major head injury
* Any brain devices/implants (including cochlear implants and aneurysm clips)
* Braids or other hair styling that prevents direct access to the scalp (if removal not possible)
* Skin allergies or very sensitive skin
* Pregnant or nursing females
* Failure to pass a urinary drug test at the first session
* Use of hormonal birth control or supplements in the past two weeks
* Non English speakers
* Cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2017-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Stimulation, Then Alpha Stimulation: Participants will receive sham stimulation at the first session. Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham. Then, participants will receive 2 mA of alternating current stimulation at a frequency of 10 Hz for 40 minutes at the first session. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator Sham: The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session.
- Alpha Stimulation, Then Sham Stimulation: Participants will receive 2 mA of alternating current stimulation at a frequency of 10 Hz for 40 minutes at the first session. tACS stimulation is delivered using the XCSITE100 Stimulator tACS. Then, participants will receive sham stimulation at the second session. Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
Period: First Session
Arm/Group | Sham Stimulation, Then Alpha Stimulation | Alpha Stimulation, Then Sham Stimulation
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period (5-9 Days)
Arm/Group | Sham Stimulation, Then Alpha Stimulation | Alpha Stimulation, Then Sham Stimulation
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Session
Arm/Group | Sham Stimulation, Then Alpha Stimulation | Alpha Stimulation, Then Sham Stimulation
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Group (Both Sham and Alpha Stimulation): Participants received sham stimulation at one session and alpha stimulation at the other in a randomized order. Sessions were separated by 5-9 days.
Arm/Group | Overall Group (Both Sham and Alpha Stimulation)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Salivary Alpha Amylase
Description: Change after stimulation
Time Frame: Before and after 40-minute stimulation at each session.
Measure: Mean (Standard Deviation); unit: log-normalized percent change of U/mL
Groups:
- Sham Stimulation: Sham Stimulation mimics the physical effects of stimulation, with up to one minute of stimulation during the session. Sham stimulation is delivered using the XCSITE100 Stimulator Sham.
  XCSITE100 Stimulator Sham: The participant will receive up to one minute of tACS stimulation until the stimulation fades. Sham stimulation mimics the skin sensations a participant would experience during a tACS session.
- Alpha Stimulation: Participants will receive 2 mA of alternating current stimulation at a frequency of 10 Hz for 40 minutes. tACS stimulation is delivered using the XCSITE100 Stimulator tACS.
  XCSITE100 Stimulator tACS: Transcranial alternating current stimulation (tACS) is a method of noninvasive brain stimulation in which weak electrical current are applied to the scalp in a sine wave pattern to induce cortical oscillations at the frequency at which they are applied.
Arm/Group | Sham Stimulation | Alpha Stimulation
Number analyzed (Participants) | 20 | 20
log-normalized percent change of U/mL | 0.00695 (0.196) | 0.03055 (0.188)
Statistical Analysis 1: Comparison: Sham Stimulation vs Alpha Stimulation; Test type: Equivalence — ANOVA; p = 0.70, ANOVA — P value threshold is 0.05

2. Primary Outcome: Salivary Cortisol
Description: Change before and after stimulation
Time Frame: Before and after 40 minutes of stimulation
Measure: Mean (Standard Deviation); unit: log-normalized percent change µg/dL
Arm/Group | Sham Stimulation | Alpha Stimulation
Number analyzed (Participants) | 20 | 20
log-normalized percent change µg/dL | -0.0551 (0.168) | -0.0702 (0.164)
Statistical Analysis 1: Comparison: Sham Stimulation vs Alpha Stimulation; Test type: Equivalence — ANOVA; p = 0.71, ANOVA — P value threshold is 0.05

3. Secondary Outcome: Heart Rate Variability
Description: Change in the ratio between the power in low frequency band and the power in high frequency band. As this outcome variable is a ratio between two items that are measured in microvolt^2, the ratio does not have a unit of measure.
Time Frame: Before and after 40-minute stimulation at each session.
Measure: Mean (Standard Deviation); unit: log-normalized percent change
Arm/Group | Sham Stimulation | Alpha Stimulation
Number analyzed (Participants) | 20 | 20
log-normalized percent change | 1.599 (3.33) | 0.308 (3.70)

4. Secondary Outcome: Percent Change in Respiration
Description: Respiration rate, measured via a belt placed around the participant's abdomen as breaths per second.
Time Frame: Before and after 40-minute stimulation at each session.
Measure: Mean (Standard Deviation); unit: Percent change in breaths per second
Arm/Group | Sham Stimulation | Alpha Stimulation
Number analyzed (Participants) | 20 | 20
Percent change in breaths per second | -0.0075 (0.076) | 0.0325 (0.093)

5. Secondary Outcome: Electroencephalogram (EEG)
Description: The investigators will compare alpha oscillation power from resting-state EEG recordings before and after stimulation/sham at each session.
Time Frame: Before and after 40-minute stimulation at each session.
Measure: Mean (Standard Deviation); unit: percent change of uV^2/Hz
Arm/Group | Sham Stimulation | Alpha Stimulation
Number analyzed (Participants) | 20 | 20
percent change of uV^2/Hz | -0.0087 (0.0360) | 0.0114 (0.0752)

ADVERSE EVENTS:
Time Frame: From first session until completion of second session for each participant, for a total of 7-11 days (including both session days and 5-9 days of washout).
Arm/Group | Sham Stimulation | Alpha Stimulation
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03178344/Prot_SAP_000.pdf